CLINICAL TRIAL: NCT03752229
Title: A Randomized, Single Blind, Uni-centre Study in Healthy Volunteers, to Determine Capillary Blood Volume and Pain Perception Obtained in a Process of Puncturing With Different Safety Lancets
Brief Title: Capillary Blood Volume and Pain Perception Obtained in a Process of Puncturing With Different Safety Lancets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 02LAN2017
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: safety lancets; lancet; capillary blood; capillary blood sampling; blood volume; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- HTL-STREFA S.A.safety lancet type 610 (Experimental)
  Interventions: Device: Acti-Lance Lite; Device: Acti-Lance Universal; Device: Acti-Lance Special
- HTL-STREFA S.A.safety lancet type 553-556 (Experimental)
  Interventions: Device: Medlance Plus Super Lite; Device: Medlance Plus Lite; Device: Medlance Plus Universal; Device: Medlance Plus Extra; Device: Medlance Plus Special
- HTL-STREFA S.A.safety lancet type 430 (Experimental)
  Interventions: Device: Prolance Micro Flow; Device: Prolance Low Flow; Device: Prolance Normal Flow; Device: Prolance High Flow; Device: Prolance Max Flow; Device: Prolance Pediatric
- HTL-STREFA S.A.safety lancet type 420 (Experimental)
  Interventions: Device: Haemolance Micro Flow; Device: Haemolance Low Flow; Device: Haemolnace Normal Flow; Device: Haemolance High Flow; Device: Haemolance Max Flow; Device: Haemolance Pediatric
- HTL-STREFA S.A.safety lancet type 520 (Experimental)
  Interventions: Device: MediSafe Solo 29 Gauge; Device: MediSafe Solo 23 Gauge
- HTL-STREFA S.A.safety lancet type 450 (Experimental)
  Interventions: Device: ergoLance Micro Flow; Device: ergoLance Normal Flow; Device: ergoLance High Flow
- HTL-STREFA S.A.safety lancet type 545-549 (Experimental)
  Interventions: Device: Medlance (light blue); Device: Medlance (blue); Device: Medlance (dark blue); Device: Medlance (yellow); Device: Medlance (orange); Device: Medlance (red)
- Owem Mumford lancet (Experimental)
  Interventions: Device: Unistik 3 Extra; Device: Unistik 3 Comfort; Device: Unistik Touch
- Medicore lancet (Experimental)
  Interventions: Device: ReadyLance (blue); Device: ReadyLance (orange)
- Arkray lancet (Experimental)
  Interventions: Device: AssureLance; Device: AssureLance MicroFlow
- Medipurpose lancet (Experimental)
  Interventions: Device: Surgilance; Device: Surgilance Lite (grey); Device: Surgilance Lite (purple)
- Sterilance lancet (Experimental)
  Interventions: Device: SteriLance Lite2; Device: SteriLance Press
- Dynarex lancet (Experimental)
  Interventions: Device: SensiLance (pink); Device: SensiLance (orange)
- Ypsomed lancet (Experimental)
  Interventions: Device: mylife
- Promismed lancet (Experimental)
  Interventions: Device: VeriFine
- Cambridge Sensors lancet (Experimental)
  Interventions: Device: Microdot

INTERVENTIONS:
Device: Acti-Lance Lite — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 610
  Arms: HTL-STREFA S.A.safety lancet type 610
Device: Acti-Lance Universal — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 610
  Arms: HTL-STREFA S.A.safety lancet type 610
Device: Acti-Lance Special — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 610
  Arms: HTL-STREFA S.A.safety lancet type 610
Device: Medlance Plus Super Lite — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 553
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Lite — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 553
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Universal — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 554
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Extra — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 555
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Medlance Plus Special — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 556
  Arms: HTL-STREFA S.A.safety lancet type 553-556
Device: Prolance Micro Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Low Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Normal Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance High Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Max Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Prolance Pediatric — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 430
  Arms: HTL-STREFA S.A.safety lancet type 430
Device: Haemolance Micro Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 420
  Arms: HTL-STREFA S.A.safety lancet type 420
Device: Haemolance Low Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 420
  Arms: HTL-STREFA S.A.safety lancet type 420
Device: Haemolnace Normal Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 420
  Arms: HTL-STREFA S.A.safety lancet type 420
Device: Haemolance High Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 420
  Arms: HTL-STREFA S.A.safety lancet type 420
Device: Haemolance Max Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 420
  Arms: HTL-STREFA S.A.safety lancet type 420
Device: Haemolance Pediatric — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 420
  Arms: HTL-STREFA S.A.safety lancet type 420
Device: MediSafe Solo 29 Gauge — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 520
  Arms: HTL-STREFA S.A.safety lancet type 520
Device: MediSafe Solo 23 Gauge — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 520
  Arms: HTL-STREFA S.A.safety lancet type 520
Device: ergoLance Micro Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 450
  Arms: HTL-STREFA S.A.safety lancet type 450
Device: ergoLance Normal Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 450
  Arms: HTL-STREFA S.A.safety lancet type 450
Device: ergoLance High Flow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 450
  Arms: HTL-STREFA S.A.safety lancet type 450
Device: Medlance (light blue) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 545
  Arms: HTL-STREFA S.A.safety lancet type 545-549
Device: Medlance (blue) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 545
  Arms: HTL-STREFA S.A.safety lancet type 545-549
Device: Medlance (dark blue) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 546
  Arms: HTL-STREFA S.A.safety lancet type 545-549
Device: Medlance (yellow) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 547
  Arms: HTL-STREFA S.A.safety lancet type 545-549
Device: Medlance (orange) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 548
  Arms: HTL-STREFA S.A.safety lancet type 545-549
Device: Medlance (red) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: HTL-STREFA S.A. safety lancet type 549
  Arms: HTL-STREFA S.A.safety lancet type 545-549
Device: Unistik 3 Extra — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Owem Mumford lancet
  Arms: Owem Mumford lancet
Device: Unistik 3 Comfort — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Owem Mumford lancet
  Arms: Owem Mumford lancet
Device: Unistik Touch — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Owem Mumford lancet
  Arms: Owem Mumford lancet
Device: ReadyLance (blue) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Medicore lancet
  Arms: Medicore lancet
Device: ReadyLance (orange) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Medicore lancet
  Arms: Medicore lancet
Device: AssureLance — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Arkray lancet
  Arms: Arkray lancet
Device: AssureLance MicroFlow — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Arkray lancet
  Arms: Arkray lancet
Device: Surgilance — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Medipurpose lancet
  Arms: Medipurpose lancet
Device: Surgilance Lite (grey) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Medipurpose lancet
  Arms: Medipurpose lancet
Device: Surgilance Lite (purple) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Medipurpose lancet
  Arms: Medipurpose lancet
Device: SteriLance Lite2 — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Sterilance lancet
  Arms: Sterilance lancet
Device: SensiLance (pink) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Dynarex lancet
  Arms: Dynarex lancet
Device: SteriLance Press — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Sterilance lancet
  Arms: Sterilance lancet
Device: SensiLance (orange) — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Dynarex lancet
  Arms: Dynarex lancet
Device: mylife — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Ypsomed lancet
  Arms: Ypsomed lancet
Device: VeriFine — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Promismed lancet
  Arms: Promismed lancet
Device: Microdot — Finger lancing was undertaken in a standardized way and was performed by medical staff trained from lancing procedure described in the Protocol.
  Total blood collection time was recorded in the source documentation and then volume of the blood was measured using a calibrated ruler.
  Other Names: Cambridge Sensors lancet
  Arms: Cambridge Sensors lancet

SUMMARY:
The study was a randomized, single blind, uni-center pivotal study in male and female healthy volunteers, to determine capillary blood volume and pain perception obtained in a process of puncturing with different safety lancets.

A group of three hundred (300) Caucasian male and female Subjects was randomized (aged > 18 to < 65 years old) who were in good physical and mental condition. The Subjects had 4 (four) fingers (two fingers from each hand) lanced each with a different type of safety lancet. Overall, 4 (four) different safety lancets were investigated per each Subject.

Overall, 48 (forty eight) different safety lancets (4 different safety lancets per one Subject) were investigated, the capillary blood volume and pain were measured.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent.
* Male and female volunteers
* Age between 18 and 65 inclusive
* Able to communicate well with the Investigator and comply with the requirements of the study
* Volunteers who are in good physical and mental health

Exclusion Criteria:

* Confirmed or suspected malignant cancer
* Pregnancy or breastfeeding (only for women with childbearing potential based on pregnancy test conducted at Site)
* History of poor blood circulation.
* Any skin condition on his or her fingers that prevents blood sampling
* Anxiety with needles or finger pricks
* Clotting disorders (including bleeding) in medical history
* Neuropathy or other condition affecting sensation in the hands.
* History of blood borne infection (e.g., HIV, hepatitis B or C, syphilis, malaria, babesiosis, brucellosis, leptospirosis, arboviral infections, relapsing fever, T lymphotropic virus Type 1, Creutzfeldt-Jakob disease)
* Currently participating in another study
* History of drug or alcohol abuse within the 12 months prior to screening or evidence of such abuse
* Intake of alcohol within 48 hours prior to the start of the study (self-reporting)
* Donation or loss of 400 mL or more of blood within 4 weeks prior to the start of the study
* Any other condition that in the Investigator opinion may negatively influence Subject's participation in the study
* Intake of medicines that affect blood coagulability (including anticoagulants such as vitamin K, antivirals and anticoagulants such as heparin, aspirin, thrombin inhibitors, vitamin K antagonists).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Volume (microliters) of blood in the capillary tube | The blood volume was noted after 20 seconds
  The amount of capillary blood volume collected after a single lancing of the fingertip.
Volume (microliters) of blood in the capillary tube | The blood volume was noted until the end of bleeding or up to 2 minutes time
  The amount of capillary blood volume collected after a single lancing of the fingertip.

SECONDARY OUTCOMES:
Pain perception | directly after lancing
  The intensity of pain perceived by the patient was assessed with the use of the numeric Visual Analog Scale (VAS). The Subject marked on the scale the number from 0 ("no pain") to 10 ("worst imaginable pain") that represented their perception of pain. A higher score indicated greater pain intensity.
Pain perception | after 30 minutes ± 5 min after lancing
  The intensity of pain perceived by the patient was assessed with the use of the numeric Visual Analog Scale (VAS). The Subject marked on the scale the number from 0 ("no pain") to 10 ("worst imaginable pain") that represented their perception of pain. A higher score indicated greater pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- BioResearch Group Sp. z o.o., Nadarzyn, Masovian Voivodeship, Poland